CLINICAL TRIAL: NCT06881953
Title: Prevention Strategy for Respiratory Syncytial Virus (RSV) Infections in Infants: Maternal Vaccination During Pregnancy or Direct Immunization of Children? A French Online Study
Brief Title: Prevention Strategy for Respiratory Syncytial Virus (RSV) Infections in Infants in France
Acronym: SPIRAV
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP250429
Record Dates: First submitted 2025-03-11; First posted 2025-03-18 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-03

CONDITIONS: RSV Infection
Keywords: Respiratory syncytial virus; nirsevimab; vaccine; health campaign
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — The questionnaire will be completed on line by the participants (approx. 10 min).

SUMMARY:
Bronchiolitis is a viral lower respiratory tract infection, caused in 50 to 80% of cases by the respiratory syncytial virus (RSV).

Although generally mild, RSV bronchiolitis remains the leading cause of infant hospitalizations for acute respiratory distress in Europe. In France, nearly 30% of children under two years of age are affected annually, representing approximately 480,000 cases. RSV bronchiolitis accounts for 2 to 3% of hospital admissions among infants under one year each winter. These situations place a significant burden on pediatric intensive care units and emergency departments, impacting the delivery of care for other pediatric patients and raising concerns among parent and families.

Until September 2023, RSV lower respiratory tract infection prevention strategies in infants in France were limited to non-pharmacological barrier measures, with a monthly injection of the monoclonal antibody palivizumab (Synagis®) recommended among high-risk infants, particularly those born preterm before 35 weeks of gestation.

At the end of 2023, a new monoclonal antibody, nirsevimab (Beyfortus®), indicated for passive immunization in the general infant population, received marketing authorization. Administered as a single dose to neonates (from birth) and infants during their first RSV season, nirsevimab demonstrated an estimated efficacy of 76% to 83% in preventing severe RSV bronchiolitis during the 2023-2024 epidemic in France. At the same time, the RSV vaccine Abrysvo® (Pfizer) became available in France since September 2024, following European marketing authorization in August 2023. Administered during the third trimester of pregnancy, this maternal immunization strategy aims to confer passive immunity to neonates (from birth up to six months of age) through transplacental transfer of RSV-specific maternal antibodies.

For the 2024-2025 RSV season, the national prevention strategy for RSV-related respiratory infections in infants is based on general non-pharmacological measures and, between September 15, 2024, and January 31, 2025, on maternal vaccination (administered between 32 and 36 weeks of gestation) and/or direct administration of nirsevimab to neonates.

To date, no population-based data are available in France regarding maternal adherence to the current RSV prevention strategy for respiratory syncytial virus (RSV) infections in infants. The acceptability of maternal RSV vaccination remains unknown, as well as the factors associated with the choice between the two recommended strategies and the reasons given by pregnant women for their decision.

The objective of this study is to assess, in population, the adherence of pregnant women to the current RSV infection prevention strategy for infants in France, which has not yet been studied. The study will focus on the method most commonly chosen by women (maternal vaccination with Abrysvo® during pregnancy or administration of nirsevimab (Beyfortus®) to their neonates), aiming to identify the factors associated with the choice of one strategy over the other and to describe the main reasons women give for their decision to either follow or not follow one of the prevention strategies.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Able to speak and understand French well enough to read and comprehend the information leaflet and the questionnaire
* Delivery in metropolitan France between October 1, 2024, and January 31, 2025
* Live-born child
* Term-born child (37 weeks of gestation or more)
* No objection to participating in the study

Exclusion Criteria:

* Women under legal protection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — as this study is concerned with pregnancy and maternity, only women will be included.
Study Population: Women who gave birth at term in metropolitan France between October 1, 2024, and January 31 or February 2025 (i.e., during the first implementation period of the RSV-related lower respiratory infection prevention strategy for infants in metropolitan France)
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-06-17 (Actual); Primary Completion 2025-12-17 (Estimated); Study Completion 2025-12-17 (Estimated)

PRIMARY OUTCOMES:
Adherence of pregnant women to the current RSV infection prevention strategy for infants in France. | Through study time period, 6 months
  The primary aim of this study is to assess the adherence of pregnant women to the current RSV infection prevention strategy for infants in France, defined as the administration of the RSV vaccine Abrysvo® during pregnancy and/or the direct administration of specific monoclonal antibodies (nirsevimab, Beyfortus®) to the neonate.

SECONDARY OUTCOMES:
Assessing the factors associated with overall adherence to this prevention strategy. | Through study time period, 6 months
  Through online questionnaire
Identifying and assessing the maternal and organizational factors associated with the choice of maternal vaccination or administration of nirsevimab to the neonate. | Through study time period, 6 months
  Through online questionnaire
Describing the main reasons reported by women to explain their decision to follow or not follow one of the prevention strategies. | Through study time period, 6 months
  Through online questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Public health department, Hôpital Pitié Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon reasonable request The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.